CLINICAL TRIAL: NCT04320121
Title: Effect of Nelutri™ on Musculoskeletal Biomarkers in Relative Sarcopenia Adults: a Randomized, Double-blinded, Placebo-controlled Trial
Brief Title: Effect of Nelutri™ on Musculoskeletal Biomarkers in Relative Sarcopenia Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Sang Yeoup Lee, Professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 02-2020-005
Record Dates: First submitted 2020-03-17; First posted 2020-03-24 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Muscular Sarcoidosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nelutri™ group (Experimental): This group takes Nelutri™ for 12 weeks
  Interventions: Dietary Supplement: Nelutri™
- Placebo group (Placebo Comparator): This group takes placebo for 12 weeks
  Interventions: Dietary Supplement: Placebo group

INTERVENTIONS:
Dietary Supplement: Nelutri™ — Nelutri™ 2,000 mg/day for 12 weeks
  Arms: Nelutri™ group
Dietary Supplement: Placebo group — Placebo 2,000 mg/day for 12 weeks
  Arms: Placebo group

SUMMARY:
The investigators conduct a randomized, double-blind, placebo-controlled study to investigate the effects of Nelutri™on muscle strength, muscle mass, and muscle function in healthy adults for 12 weeks.

DETAILED DESCRIPTION:
A previous study has indicated that Nelutri™ may increase muscle mass and strength. Therefore, the investigators conduct a randomized, double-blind, placebo-controlled study to investigate the effects of Nelutri™on muscle strength, muscle mass, and muscle function in healthy adults; the safety of the compound are also evaluate. The Investigators examine the peak torque/body weight at 60°/s knee extension, handgrip strength, skeletal muscle mass, physical performance, and metabolic parameters at baseline, as well as after 6 and 12 weeks of intervention. Eighty adults were administered either 2,000 mg of Nelutri™ or a placebo each day for 12 weeks;

ELIGIBILITY:
Inclusion Criteria:

* <110% of the standard lean body mass as measured using the body composition analyzer
* Body-mass index (BMI) ranging from 18.5 to 30.0 kg/m2
* Those who have an average protein intake of 60 g or more/day.

Exclusion Criteria:

* Abnormal liver or renal function (i.e., serum aminotransferase activity > 60 IU/L and serum creatinine concentrations > 1.2 mg/dL)
* Diabetes (diagnosed clinically or fasting glucose level > 126 mg/dL)
* History of fracture during the previous year
* Uncontrolled hypertension
* History of serious cardiac disease such as angina or myocardial infarction
* History of gastrectomy
* History of medication for psychiatric disease
* Administration of oriental medicine including herbs within the past 4 weeks
* Evidence of relatively high skeletal mass (more than 110% of the standard lean body mass as measured using the body composition analyzer

Min Age: 19 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
muscle strength | 12 weeks
  the peak torque at 60°/s knee extension (/kg)

SECONDARY OUTCOMES:
appendicular skeletal mass/(height x height) | 12 weeks
  using dual-energy X-ray absorptiometry
appendicular skeletal mass/weight x 100 | 12 weeks
  using dual-energy X-ray absorptiometry
Skeletal Muscle Mass Index/(height x height) | 12 weeks
  using dual-energy X-ray absorptiometry
Creatinine Kinase | 12 weeks
  Creatinine Kinase
Lactate | 12 weeks
  Lactate
EuroQol five dimensional three levels (EQ-5D-3L) | 12 weeks
  an index of life quality, minimum, maximum values (-0.171, 1), higher scores mean a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Sang Yeoup Lee, MD, Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, Gyeungsangnam-do, South Korea

IPD SHARING:
Plan to Share IPD: No